CLINICAL TRIAL: NCT00518544
Title: Hemostatic Effect of Various Colloid Solutions According to Blood Types
Brief Title: Hemostatic Effect of Various Colloid Solutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRS107-17-1
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Laminectomy
Keywords: hydroxyethyl starch, blood type, coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: administration of hydroxyehtyl starch — colloid is administered during operation according to blood loss.

SUMMARY:
Background: Individuals with type O blood have reduced factor VIII and von Willebrand factor levels compared to the non-O counterpart. Infusion of hydroxyethyl starch (HES) impairs coagulation and, in O blood type, apparent coagulopathy can develop after HES infusion. A newly market-released balanced HES (670/0.75) has physiologic pH and balanced electrolytes including calcium, which are beneficial to coagulation. Studies comparing balanced HES (670/0.75) with saline-based HES (130/0.4), previously known the least coagulopathic are rare. Therefore, we try to reveal the difference of coagulation, pH/electrolyte balance, and bleeding amount between the non-O and O blood types after infusion of these two newest HES.

Methods: Each 20 of non-O and type O ASA 1 or 2 patients scheduled for spinal surgery involving 2 or 3 spinal levels were enrolled. 20 ml/kg of saline-based HES (130/0.4) or balanced HES (670/0.75) was administered during operation. Blood loss, coagulation and metabolic profiles were checked at pre-infusion (T0), 5 min after infusion (T1), 4 hrs after infusion (T2) and 24 hrs after infusion (T4).

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA 1 or 2, and scheduled for posterior laminectomy and internal fixation at two or three spinal levels.

Exclusion Criteria:

* the presence of cardiovascular diseases, cerebral vascular disease, hepatic, pulmonary, or renal disease, hemoglobin < 12 g/dl, platelet count < 150,000 /ml, coagulopathy, taking medication likely to alter coagulation less than 2 weeks before the study, or an allergic reaction to HES

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-07

PRIMARY OUTCOMES:
Blood loss, coagulation and metabolic profiles | pre-infusion, 5 min after infusion, 4 hrs after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, MD., PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea